CLINICAL TRIAL: NCT00960700
Title: Clinical Investigational Plan of the Rayner M-flex Multifocal Intraocular Lens (IOL) With Different Near Additions
Brief Title: A Multi Focal Visual Outcome Study Using Different Near Additions
Status: Terminated | Type: Observational
Sponsor: Rayner Intraocular Lenses Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: Rayner-630F
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Cataract; Aphakia
Keywords: MFlex; Multifocal; 630F
MeSH Terms: conditions — Cataract; Aphakia | interventions — Visual Acuity; Contrast Sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Visual Acuity — Assessment of visual acuity
Device: Contrast sensitivity — Assessment of contrast sensitivity
Device: Reading Speed — Assessment of reading speed
Procedure: Eye Health — Examination of eye health through use of a slitlamp/ photography. Assessment of Intraocular Pressure.

SUMMARY:
A multi-centre non-randomized clinical investigation to assess multifocal visual outcomes using different near additions, for the treatment of aphakia after cataract removal.

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract patients undergoing cataract surgery where the cataractous lens has been removed by phacoemulsification, with circular tear capsulotomy, leaving the posterior capsule intact
* Patients requiring primary IOL implantation
* Patients with a potential corrected visual acuity of 20/40 or better on clinical assessment
* Patients with normal anterior segments - apart from cataracts
* Subjects with clear intraocular media other than cataract

Exclusion Criteria:

* Pre-existing pathology or physiology, which may be aggravated by the implant, or may render the implant ineffective and that could potentially cause future acuity losses to a level of 0.5 or 20/40 or worse in either eye. This includes the following:

  * Microphthalmia
  * Corneal decompensation or Endothelial Insufficiency
  * Pseudo exfoliation
  * High myopia
  * Pars planitis
* Patient with greater than 1 dioptre of pre-operative corneal astigmatism
* Subjects who are expected to require retinal laser treatment
* Previous intraocular and/or corneal surgery
* History of uveitis, glaucoma, proliferative diabetic retinopathy or IDDM, pseudoexfoliation, macular degeneration that may affect potential best corrected visual acuity of 20/40 or better
* Operative complications of posterior capsular rupture, zonular dehiscence, incomplete continuous curvilinear capsulorhexis, severe iris /corneal trauma and inability to achieve secure placement in the designated location
* Subjects using a systemic medication that is known to cause ocular side effects
* Subjects participating in a concurrent clinical trial or if they have participated in an ophthalmology clinical trial within the last 30 days
* Subjects who have only one eye with potentially good vision
* Patients who are not willing to cooperate in the 6-months follow-up period
* Children under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aphakic adults with potential for > 20/40 visual outcome to participate in a binocular study. Subjects to be implanted bilaterally with study device.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Visual acuity at distance and near | 1 year

SECONDARY OUTCOMES:
Range of clear vision | 1 year
Reading speed | 1 year
Cntrast sensitivity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Gerd U Auffarth, Prof., Principal Investigator
Locations (2):
- Ruprecht- Karl Universitat Heidelberg, Abteilung Augenheilkunde, Heidelberg, Germany
- Eye Clinic and national Centre of Ophthalmology, Kaunas, Lithuania

REFERENCES:
- See also: Publication from the results — http://www.ncbi.nlm.nih.gov/pubmed/23290317